CLINICAL TRIAL: NCT01659385
Title: Assessment of Serum Leptin Levels in Females With Papillary Thyroid Carcinoma, Benign Thyroid Nodules, and Normal Controls
Brief Title: Leptin Levels in Papillary Thyroid Cancer
Acronym: LL-PTC
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0276-12-EP
Record Dates: First submitted 2012-08-03; First posted 2012-08-07 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Thyroid Cancer, Papillary; Leptin Levels
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate Leptin levels in females, in the setting of papillary thyroid cancer, benign thyroid nodules, and in normal females without thyroid disease.

DETAILED DESCRIPTION:
There will be three groups in this study, but 2 of the groups are part of another study so will only recruit normal controls.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age>/- 19
* Not currently pregnant or lactating
* Normal thyroid gland by history

Exclusion Criteria:

* Male Gender
* Pregnancy
* Lactation
* Age below 19
* Abnormal thyroid gland by history
* Abnormal thyroid gland by structure using ultrasound
* Abnormal thyroid gland by function using TSH, Free T4

Ages: 19 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Females with no prior history of thyroid disease and not on thyroid medications.
  Active recruitment will be for normal controls only. They will be age and weight/height matched to females with prior diagnosis of thyroid cancer or thyroid nodules who are already part of another study.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2012-08-07 (Actual); Primary Completion 2013-04-25 (Actual); Study Completion 2013-04-25 (Actual)

PRIMARY OUTCOMES:
evaluating Leptin level Evaluating Serum Leptin Levels Between 3 Groups. One Group with Papillary Thyroid Carcinoma. One Group With Benign Nodules. One Group with Normal Thyroid. | During Study
  Assessing serum leptin levels in females with treated papillary thyroid carcinoma and compared to females with proven benign thyroid nodules and females with normal thyroid glands. All groups were matched by gender, age, and BMI to limit confounders.

CONTACTS AND LOCATIONS:
Overall Officials: Whitney Goldner, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States